CLINICAL TRIAL: NCT00555594
Title: Prospective Study to Determine the Effect of Subconjunctival Bevacizumab (AVASTIN) in Corneal Neovascularization
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Collaborators: National Council of Science and Technology, Mexico (Other); Universidad Nacional Autonoma de Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cornea2
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Corneal Neovascularization
Keywords: corneal neovascularization; Bevacizumab (Avastin); Immunologic rejection; vascular endothelial growth factor
MeSH Terms: conditions — Corneal Neovascularization | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Patients with corneal neovascularization of infectious etiology, steroid reactors, and know glaucoma or glaucoma suspects. They received one dose of 0.1cc of subconjunctival Bevacizumab (Avastin™ Genentech, Inc, USA) in bulbar conjunctiva, 2 mm from the limbus, according to the location of the vessels.
  Interventions: Drug: Bevacizumab (Avastin)
- B (Active Comparator): Patients with corneal neovascularization of any cause except for infectious disease. Patients of this group received one application of 0.1cc of subconjunctival Bevacizumab™ + 0.1cc of triamcinolone acetonide (ATLC; Grin laboratories, México city) in bulbar conjunctiva, 2 mm from de limbus, according to the location of the vessels.
  Interventions: Drug: Bevacizumab (Avastin)

INTERVENTIONS:
Drug: Bevacizumab (Avastin) — One dose of 0.1cc of subconjunctival Bevacizumab was applied

SUMMARY:
To determine the effect of subconjunctival Bevacizumab in corneal neovascularization

DETAILED DESCRIPTION:
Corneal transplantation is the most commonly performed transplant surgery in the world today. Immunologic rejection is the leading cause of graft failure, with about 25% of graft recipients experiencing at least one episode of rejection. Of these episodes, about 20% are irreversible. The rate of corneal graft rejection in high-risk eyes, such as corneal neovascularization, has been reported to be 50% to 70%. Vascularized corneas have a much higher rate of graft rejection than avascular corneas. Whereas the normal cornea is devoid of blood and lymphatic vessels, both can invade the cornea secondary to a variety of corneal diseases and after surgery. This not only reduces visual acuity, but also renders such a cornea high-risk, if subsequent corneal transplantation is performed.Anti-angiogenesis, the pharmacologic inhibition of new blood vessel growth and formation, is a new treatment strategy under active and vigorous investigation. Multiple growth factors have been shown to contribute to the molecular events involved in the regulation of blood vessel growth Similarly, it is assumed that angiogenic growth factors such as vascular endothelial growth factor (VEGF), considered a major pro-angiogenic factor, could play a role in the pathogenesis of neovascularization.

Several approaches can be taken to neutralize VEGF. Bevacizumab (Avastin) is a full-length humanized murine monoclonal antibody against the VEGF molecule.It binds to and inhibits the biologic activity of human VEGF preventing the interaction of this molecule to its receptors on the surface of endothelial cells. The interaction of VEGF with its receptors leads to endothelial cell proliferation and new vessel formation.

There is evidence that triamcinolone acetonide (TA) inhibits vasogenic edema and inflammation, decreases vascular leakage, reduces the secretion of VEGF by pigment epithelial cells during oxidative stress and, down-regulates the expression of the VEGF gene in vascular smooth muscle cells Furthermore, TA decreases the paracellular permeability of cultured epithelial cells and down-regulates the inflammatory expression of endothelial adhesion molecules.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of vessels in minimum one quadrant
2. vessels that penetrate more than 0.5 mm of the limb, in any depth
3. who had signed the informed consent
4. those that could attend to frequent ophthalmologic revisions after treatment and could wait for 6 months before the surgical procedure.

Exclusion Criteria:

1. Patients with urgent need of a penetrating keratoplasty, pregnancy or lactancy
2. Patient that may need an additional procedure to penetrating keratoplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2006-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Anterior segment slit-lamp photographs and fluorescein angiograms Compared for any sign of diminished vascularization | three weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hernández-Quintela Everardo, MD, Principal Investigator — Consejo Nacional de Ciencia y Tecnología (CONACYT) grant no. 115755 (EHQ)
Locations (1):
- Asociación Para Evitar la Ceguera en México, IAP, Hospital "Dr. Luis Sánchez Bulnes", Mexico City, Mexico

REFERENCES:
- [Background] Foulks GN, Sanfilippo FP, Locascio JA 3rd, MacQueen JM, Dawson DV. Histocompatibility testing for keratoplasty in high-risk patients. Ophthalmology. 1983 Mar;90(3):239-44. doi: 10.1016/s0161-6420(83)34575-9. PMID 6346199
- [Background] Cursiefen C, Seitz B, Dana MR, Streilein JW. [Angiogenesis and lymphangiogenesis in the cornea. Pathogenesis, clinical implications and treatment options]. Ophthalmologe. 2003 Apr;100(4):292-9. doi: 10.1007/s00347-003-0798-y. German. PMID 12682761
- [Background] Ciardella AP, Donsoff IM, Guyer DR, Adamis A, Yannuzzi LA. Antiangiogenesis agents. Ophthalmol Clin North Am. 2002 Dec;15(4):453-8. doi: 10.1016/s0896-1549(02)00042-1. PMID 12515077
- [Background] Foulks GN, Sanfilippo F. Beneficial effects of histocompatibility in high-risk corneal transplantation. Am J Ophthalmol. 1982 Nov;94(5):622-9. doi: 10.1016/0002-9394(82)90007-1. PMID 6756156
- [Background] Norrby K. In vivo models of angiogenesis. J Cell Mol Med. 2006 Jul-Sep;10(3):588-612. doi: 10.1111/j.1582-4934.2006.tb00423.x. PMID 16989723
- [Background] Kuwano M, Fukushi J, Okamoto M, Nishie A, Goto H, Ishibashi T, Ono M. Angiogenesis factors. Intern Med. 2001 Jul;40(7):565-72. doi: 10.2169/internalmedicine.40.565. PMID 11506294
- [Background] Kvanta A, Sarman S, Fagerholm P, Seregard S, Steen B. Expression of matrix metalloproteinase-2 (MMP-2) and vascular endothelial growth factor (VEGF) in inflammation-associated corneal neovascularization. Exp Eye Res. 2000 Apr;70(4):419-28. doi: 10.1006/exer.1999.0790. PMID 10865990
- [Background] Gan L, Fagerholm P, Palmblad J. Vascular endothelial growth factor (VEGF) and its receptor VEGFR-2 in the regulation of corneal neovascularization and wound healing. Acta Ophthalmol Scand. 2004 Oct;82(5):557-63. doi: 10.1111/j.1600-0420.2004.00312.x. PMID 15453853
- [Background] Manzano RP, Peyman GA, Khan P, Carvounis PE, Kivilcim M, Ren M, Lake JC, Chevez-Barrios P. Inhibition of experimental corneal neovascularisation by bevacizumab (Avastin). Br J Ophthalmol. 2007 Jun;91(6):804-7. doi: 10.1136/bjo.2006.107912. Epub 2006 Dec 19. PMID 17179168
- [Background] Presta LG, Chen H, O'Connor SJ, Chisholm V, Meng YG, Krummen L, Winkler M, Ferrara N. Humanization of an anti-vascular endothelial growth factor monoclonal antibody for the therapy of solid tumors and other disorders. Cancer Res. 1997 Oct 15;57(20):4593-9. PMID 9377574